CLINICAL TRIAL: NCT05881759
Title: Integrating Food Rx With Best Feeding Practices for Chronic Disease Prevention Among EFNEP Participants
Brief Title: Integrating Food Rx With Best Feeding Practices With EFNEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Prairie View A&M University (Other); University of Houston (Other)
Responsible Party: Principal Investigator, Jayna Dave, Associate Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-50824
Record Dates: First submitted 2023-04-13; First posted 2023-05-31 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Dietary Habits; Childhood Obesity; Food Selection; Feeding Behavior
MeSH Terms: conditions — Feeding Behavior; Pediatric Obesity; Food Preferences

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Practice - ESBA (No Intervention): The control group sites will receive the existing ESBA curriculum which is their usual practice.
- ESBA + Feeding Practices (Experimental): The intervention site staff will implement the ESBA-FFYF feeding curriculum in classes using standardized implementation protocols.
  Interventions: Behavioral: Revised ESBA

INTERVENTIONS:
Behavioral: Revised ESBA — Four intervention site staff will implement the ESBA-FFYF feeding curriculum in classes using standardized implementation protocols. Two of the four intervention sites will also participate in the Food Rx program. The control group sites will receive the existing ESBA curriculum. All program materials will be available in English and Spanish. Study participation will be maintained via weekly phone calls/text messaging by the Extension staff. For the online feeding practices content, participants will receive messages to visit the project website and watch the videos, participate in online activities, and engage in facilitated online discussions. For the Food Rx arm, participants will receive a 'Food Rx' card for bi-weekly redemption of ~30 lbs of fresh produce, plus whole grains, lean protein and low-fat dairy at a co-located Houston Food Bank food pantry. The prescription will be eligible for redemption every two weeks for 3 months, for a total of 6 redemptions.
  Arms: ESBA + Feeding Practices

SUMMARY:
To assess feasibility and acceptability of of integrating Food Rx and Best Feeding Practices with EFNEP participants via a pilot study.

DETAILED DESCRIPTION:
The purpose of the pilot study is to test the FFYF feeding curriculum material and procedures for implementation, staff training, recruitment, and data collection.

ELIGIBILITY:
Inclusion Criteria:

* Living in Harris or Fort Bend counties
* being a parent of a child 4-8 years old
* ability to speak in English or Spanish
* have ready access to a telephone
* have access to the Internet with a smart phone, a tablet, a laptop, or a desktop computer

Exclusion Criteria:

* parents of children with disabilities and/or those on prescription medications that affect weight and/or appetite
* parents who are not able to complete self-report questionnaires

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in feeding practices at 3-months will be assessed using the Food Parenting Inventory | baseline and post-intervention at 3-months
  Feeding practices will be assessed using the Food Parenting Inventory

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No